CLINICAL TRIAL: NCT06217211
Title: Assessment of Ventilatory Efficacy in Patients With Fatigue Associated With SARS-CoV2 Infection After Ingestion of Beet Juice
Brief Title: Eficacia Ventilatoria y Remolacha
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Mataró (Other)
Responsible Party: Principal Investigator, Eulogio Pleguezuelos, MD PhD, Hospital de Mataró
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CEIM15/23
Record Dates: First submitted 2023-12-22; First posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: SARS CoV 2 Infection; Muscle Disorder; Fatigue
MeSH Terms: conditions — COVID-19; Muscular Diseases; Fatigue

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remolacha (Experimental): beet juice
  Interventions: Dietary Supplement: Remolacha
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Remolacha

INTERVENTIONS:
Dietary Supplement: Remolacha — BJ or PL will be administered 3 h before the start of the NO2- evaluation test since the peak in blood occurs 2-3 h after ingesting NO3-. Both drinks (BJ and PL) will be provided in an unlabeled 140ml maroon red plastic bottle. Participants will receive a randomly assigned bottle. containing 140 ml (~ 12.8 mmol, ~ 808 mg NO3-) of BJ Beet-It-Pro Elite Shot concentrate (Beet IT; James White Drinks Ltd., Ipswich, United Kingdom) or PL.

SUMMARY:
The lung is the organ most affected by COVID-19. There are patients who successfully overcome the acute COVID-19 infection and their lungs return to a normal state. However, a significant number present dyspnea and fatigue as sequelae without having a pulmonary origin, but with a significant impact on functionality. In our published studies in relation to fatigue in patients with symptoms attributed to persistent COVID, the investigators have shown that there is muscle involvement, observing a decrease in mechanical efficiency. This muscle involvement causes stimulation of ventilation through the ergoreceptors, causing ineffective ventilation. This affectation can be explained by the findings obtained in the muscle biopsies that the investigators have performed, where the investigators observed a splitting of the basement membrane of the capillaries causing an alteration in the diffusion of metabolic substrates and oxygen.

The main objective of our project is to be able to observe the response in ventilatory efficiency in patients with symptoms of post-covid fatigue after ingesting beet juice.

DETAILED DESCRIPTION:
Long COVID is a multisystem condition that comprises a set of symptoms following a SARS-CoV-2 infection. At least 65 million people around the world present symptoms associated with persistent COVID, an incidence of 10% of infected people is estimated1. The incidence is estimated at 10-30% of non-hospitalized cases, 50-70% of hospitalized cases2,3, and 10-12% of vaccinated cases4,5. Persistent COVID is associated with all ages and severity of illness in the acute phase, with the highest percentage of diagnoses between the ages of 36 and 50 years, and the majority of cases of persistent COVID are found in non-hospitalized patients with a mild acute illness6, as this population represents the majority of overall COVID-19 cases. The most prevalent symptoms in persistent COVID are fatigue, dyspnea and weakness7.

In our first published study the investigators observed that patients with fatigue after SARS CoA2 infection behaved very similarly to COPD patients, observing a decrease in mechanical efficiency (ME) at the first threshold, second threshold and at maximum consumption. of oxygen during an incremental test8. (Figure 1).

Mechanical efficiency (ME) refers to the ability of an individual to transform oxygen consumption into effective work. In other words, poorer efficiency will increase the percentage of maximum oxygen uptake (VO2max) needed to sustain a given mechanical work. A decrease in ME, indicating that more energy is expended in a given work output, could represent an increased energy cost of respiration during exercise, an altered efficiency in ATP production (ATP produced per O2 consumed), or a higher ATP cost of contraction (ATP consumed by work production)9. Patients with a decreased ME would decrease their performance and, therefore, could be limited in terms of physical activity9.

In our second study, the investigators observed that patients recovered from SARS-CoV-2 but with symptoms of fatigue presented significant muscle dysfunction compared to healthy women with similar characteristics. These findings were corroborated by detecting an increase in VO2sc and a deterioration in ME and ventilatory efficiency during the constant load test10. These results guide us towards a problem of oxygen diffusion in the muscle cell that the investigators are confirming with the findings currently obtained in quadriceps muscle biopsies. The hypothesis of causing an increase in the dilation of muscle capillaries to improve oxygen diffusion made us think about the vasodilator and ergogenic effects of beets.

Beet juice (BRJ) has become increasingly popular among athletes looking to improve sports performance. BRJ contains high concentrations of nitrate, which can be converted to nitric oxide (NO) after consumption. NO has several functions in the human body, including a vasodilatory effect, which reduces blood pressure and increases the delivery of oxygen and nutrients to various organs. BRJ consumption also has an impact on oxygen delivery to skeletal muscles, muscle efficiency, tolerance and endurance and can therefore have a positive impact on sports performance12.

Once ingested, NO3- is reduced to nitrite (NO2-) by anaerobic bacteria in the oral cavity through the action of nitrate reductase enzymes13 and then to nitric oxide (NO) in the stomach14. This physiological mechanism depends on the entero-salivary circulation of inorganic nitrate without involving the activity of NOS. Once in the stomach (at an acidic pH), nitrite is instantly decomposed to become NO and other nitrogen oxides that perform crucial physiological functions. The remaining nitrate and nitrite are absorbed from the intestine into the circulation, which can be converted to bioactive NO in tissues and blood under conditions of physiological hypoxia14. NO induces several physiological mechanisms that influence O2 utilization during contraction of the intestine. skeletal muscle. The physiological mechanisms for NO2- reduction are facilitated by hypoxic conditions, therefore NO is produced in those parts of the muscle that consume or need more O2. This mechanism would allow local blood flow to adapt to the O2 requirement, providing an adequate homogeneous distribution within the skeletal muscle. This physiological response could be positive in terms of muscle function, although it would not explain the reduction in O2 expenditure during exercise15. Another probable mechanism is related to NO2- and NO as regulators of cellular O2 utilization15.

ELIGIBILITY:
Inclusion Criteria:

* Patients with fatigue after SARS CoV2 infection.
* Written informed consent signed by the study candidates (see Addendum 1), after receiving complete information about the objectives, techniques and possible consequences of the study.

Exclusion Criteria:

* Previous cardiovascular, oncological, neuromuscular or metabolic pathologies that could interfere with the results.
* Significant alcoholism (>80 g/day) or severe malnutrition
* Chronic treatment with drugs with potential effects on muscle structure and function
* Patient treated with nitrates
* Patients diagnosed prior to the infection with fibromyalgia or chronic fatigue.
* Patient who has a contraindication to carrying out a stress test.
* Patients allergic to beets

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-11-13 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
VO2max | 1 determination per week for 3 weeks
  maximum oxygen consumption
CMT | 1 determination per week for 3 weeks
  Maximum Tolerated Load

CONTACTS AND LOCATIONS:
Locations (1):
- Eulogio Pleguezuelos, Mataró, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No